CLINICAL TRIAL: NCT02440555
Title: Evaluation of the Targeted Screening of Type 2 Diabetes by Capillary Blood Glucose Compared to Current Screening in the Priority Health Area of Saint-Etienne and the Sainté Diabète Network.
Brief Title: Evaluation of the Targeted Screening of Type 2 Diabetes by Capillary Blood Glucose
Acronym: Sainté Diabète
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS2014-2
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes, capillary blood glucose, self-administered questionnaire
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients included: fulfill the self-administered questionnaire.
  Interventions: Other: fulfill the self-administered questionnaire

INTERVENTIONS:
Other: fulfill the self-administered questionnaire — Patients viewed in a pharmacy or a hospital fulfill the self-administered questionnaire before having a capillary blood glucose measurement.

SUMMARY:
Type 2 diabetes is the chronic disease with the most important development in France, and particularly in the Saint-Etienne area due to his specific population.

Different studies showed the interest of screening targeted on high risk population to reduce cardiovascular risks and mortality.

The current screening recommandation is an opportunist targeted screening on population older than 45 years with risk factors by a fasting glucose every 3 years, and a communautaire screening targeted on population older than 45 years suffering precarity with or without risk factors by capillary blood glucose or fasting glucose.

The objective of the Sainté Diabete network is to optimize the screening of diabetics, their follow-up and their treatments. Using a self-administered questionnaire during a medical visit could be a simple, cheap and efficient tool to detect diabetics as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* 45 years or older
* Signed informed consent

Exclusion Criteria:

* fasting glucose performed in the last 2 years
* diabetes history
* not living in Saint-Etienne

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population is composed by patients living in the Saint-Etienne area, 45 years or older, not known as diabetics, and viewed in a pharmacy or a hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1305 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity of detection of type 2 diabetes | Day 1 (inclusion day)
  To evaluate the sensitivity (true positive) of detection of type 2 diabetes by a self-administered questionnaire performed in a pharmacy or a hospital compared to capillary blood glucose measurements in the same population from the priority health area of Saint-Etienne.

SECONDARY OUTCOMES:
Specificity of detection of type 2 diabetes | Day 1 (inclusion day)
  To evaluate the specificity (true negative) of detection of type 2 diabetes by a self-administered questionnaire performed in a pharmacy or a hospital compared to capillary blood glucose measurements in the same population from the priority health area of Saint-Etienne
To evaluate the cost of the targeted screening and the screening accessibility to population from the priority health area of Saint-Etienne | Month 2
To evaluate the numbers of patients screened by self-administered questionnaire and diagnosed as diabetics using fasting glucose. | Month 2

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BOIS, Pr, Study Director — Université de Saint-Etienne
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France